CLINICAL TRIAL: NCT00923338
Title: Clinical Evaluation of the Surgisis Biodesign Vesico-Vaginal Fistula Plug
Acronym: VVP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-006; 350012
Record Dates: First submitted 2009-06-16; First posted 2009-06-18 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2012-07

CONDITIONS: Vesico-vaginal Fistula
Keywords: fistula; vesico-vaginal fistula
MeSH Terms: conditions — Vesicovaginal Fistula; Fistula

ARMS (1):
- Vesico-vaginal fistula plug (Experimental): Vesico-vaginal fistula plug
  Interventions: Device: Surgisis Biodesign (Vesico-vaginal fistula plug)

INTERVENTIONS:
Device: Surgisis Biodesign (Vesico-vaginal fistula plug) — Vesico-vaginal fistula plug
  Other Names: SurgiSIS Biodesign

SUMMARY:
This clinical trial will study the safety and effectiveness of the Biodesign Vesico-vaginal fistula plug in the treatment of vesico-vaginal fistulas resulting from childbirth trauma.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed and dated the informed consent.
* Patient is 18 years old; or is an emancipated minor as defined by Ugandan law or is under 18 but has a parent/guardian who provides informed consent.
* Patient agrees to follow-up schedule.
* Patient presents with a leaking vesico-vaginal fistula, confirmed by exam, with no signs of acute inflammation, no signs of active urinary tract infection that cannot be controlled with a standard pre-operative course of antibiotics, no signs of vaginal infection, or no signs of abscess.
* Patient presents with a fistula of a size and in a location that may be reasonably treated with the VVP device.

Exclusion Criteria:

* Patient is not medically fit enough for surgery under general or spinal anesthesia.
* Patient is a "mature minor" as defined by Ugandan law.
* Patient is pregnant, breastfeeding or planning further pregnancy during the study period.
* Patient has physical allergies or cultural objections to the receipt of porcine products.
* Patient has an active sexually transmitted disease, is HIV-positive, or any other active systemic infection that may interfere with healing.
* Patient has spina bifida or other neural tube defect.
* Patient has interstitial cystitis or other chronic pelvic pain syndrome.
* Patient has signs of acute or chronic pelvic inflammation, active urinary tract infection not responsive to antibiotic treatment, vaginal infection, or abscess of the fistula tract.
* Patient presents with clinically diagnosed sepsis (for whatever reason).
* Patient has concomitant ureterovaginal fistula.

Min Age: 10 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Fistula | 4 months
Adverse Events | 4 months

SECONDARY OUTCOMES:
Improvement in quality of life | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Musa Kayondo, MD, Principal Investigator — Mbarara University Teaching Hospital
Locations (1):
- Mbarara University Teaching Hospital, Mbarara, Uganda